CLINICAL TRIAL: NCT04345263
Title: Outcome of Full Pulpotomy in Permanent Teeth With Carious Pulp Exposure, a Randomized Clinical Trial
Brief Title: Outcome of Full Pulpotomy Using Calcium Silicate Based Materials
Acronym: pulpotomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 503/2017
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Carious Teeth
Keywords: teeth, caries, pulpotomy, MTA, biodentine, bioceramic
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patient unaware of the material to be used, care provider will be given the material after performing full pulpotomy . Tooth crown will be masked during assessment of radiographs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MTA pulpotomy (Active Comparator): Tooth will receive MTA & resin composite restoration
  Interventions: Procedure: MTA pulpotomy
- Biodentine pulpotomy (Active Comparator): Tooth will receive Biodentine & resin composite restoration
  Interventions: Procedure: MTA pulpotomy
- Bioceramic pulpotomy (Active Comparator): Tooth will receive Bioceramic & resin composite restoration
  Interventions: Procedure: MTA pulpotomy

INTERVENTIONS:
Procedure: MTA pulpotomy — Cutting the coronal portion of the pulp to the level of canal orifices and applying the dressing and restoration
  Other Names: Biodentine pulpotomy and Bioceramic pulpotomy

SUMMARY:
Permanent teeth with carious pulp exposure and indicated for full pulpotomy will be treated using three different materials using aseptic technique and will be subsequently followed up clinically and radiographically at 6 months, 1 year and yearly up to 5 years.

DETAILED DESCRIPTION:
* The target sample size is 150 patients medically fit, having vital teeth with carious pulp exposure and complaining of pain.
* The patients tooth will receive full pulpotomy under aseptic conditions and it will be randomly assigned to one of 3 calcium silicate based materials namely, (Mineral trioxide Aggregate (MTA), Biodentine, and Bioceramic for capping the full pulpotomy followed by resin composite restoration.
* Follow up for pain levels will be done during the first week.
* clinical and radiographic examination will be done at 6 months, 1 year and yearly up to 5 years.
* Success of the procedure includes absence of clinical signs and symptoms, with absence of pathology in the root and periapex on periapical radiographs.
* The 3 materials will be compared in terms of clinical and radiographic outcomes.
* demographic data of the three groups will be also compared
* predictive factors of success will be also analyzed
* tooth color changes will be also measured using vita easy shade and will compared between the groups at 6 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Mature permanent tooth with carious lesion exposing the pulp,
* Positive response to cold test
* Clinical Diagnosis of reversible or irreversible pulpitis
* Restorable tooth by direct restoration or crown
* Healthy patient

Exclusion Criteria:

* Non vital teeth
* Teeth without pulp exposure
* Inability to achieve hemostasis within 10 min after pulpotomy
* Non restorable teeth or teeth that require post and core restoration

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2024-05-02 (Estimated)

PRIMARY OUTCOMES:
Degree of pain relief after treatment compared to preoperative pain level | 1 week
  Absence of symptoms or significant pain reduction within the first week after treatment as measured on a numerical scale from 0 to 10 where zero means no pain and 10 is the most sever pain. Visual analogue scale will be also used.

SECONDARY OUTCOMES:
Radiographic normalcy | 1 year and yearly up to 5 years
  Absence of pathology in the root and the bone surrounding the apex

CONTACTS AND LOCATIONS:
Overall Officials: Nessrin Taha, DCD, Study Chair — Jordan University of Science and Technology
Locations (2):
- Jordan (2):
  - Dental teaching centre Faculty Of Dentistry, Irbid
  - Jordan University of science and technology, Irbid

IPD SHARING:
Plan to Share IPD: No
Detailed participants data will be released within the publications resulting from the trial with reference to the registration number of the study. If further details are required the principal investigator. can be contacted via email.

REFERENCES:
- [Derived] Taha NA, Al-Rawash MH, Imran ZA. Outcome of full pulpotomy in mature permanent molars using 3 calcium silicate-based materials: A parallel, double blind, randomized controlled trial. Int Endod J. 2022 May;55(5):416-429. doi: 10.1111/iej.13707. Epub 2022 Mar 17. PMID 35152464